CLINICAL TRIAL: NCT03844113
Title: Carnosine for Peripheral Vascular Disease
Acronym: Car-PVD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash University (Other)
Collaborators: Monash Health (Other)
Responsible Party: Principal Investigator, Barbora de Courten, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Car-PVD
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Peripheral Arterial Disease
Keywords: carnosine; peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Carnosine

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Each participant will be given a daily oral dose 2 g of carnosine for 6 months
  Interventions: Drug: Carnosine
- Control (Placebo Comparator): Each participant will be given a daily oral dose 2 g of placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carnosine — Each participant will be given a daily oral dose 2 g of carnosine for 6 months
  Other Names: Pure Carnosine
  Arms: Intervention
Drug: Placebo — Each participant will be given a daily oral dose 2 g of methycellulose powder for 6 months
  Arms: Control

SUMMARY:
The investigators hypothesise that a home-based standardised exercise intervention with 2g of carnosine daily for 6 months will improve walking endurance in 104 patients with PVD aged 40-80 years compared to placebo and exercise through stabilisation of HIF1-α in the ischaemic leg.

Aims

Aim 1: Determine whether in patients with PVD, carnosine in addition to exercise improves:

1. walking endurance (6-min walk test; primary outcome);
2. initial claudication distance (ICD), and absolute claudication distance (ACD; treadmill), cadence, resting and exercise ABI; and
3. central blood pressure, endothelial function, arterial (aortic) stiffness, lipid profile; and
4. quality of life as determined by EuroQol-5D (all secondary outcomes).
5. Improve cognitive function (global cognitive score formed by a composite of 7 cognitive tests)

Aim 2: Delineate the mechanisms by which carnosine improves walking endurance:

1. protein expression of pro-angiogenic and carnosine related genes, including carnosine transporters in the skeletal muscle biopsies, EPCs in peripheral blood and quantitative proteomic studies.
2. other mechanisms demonstrated in animal studies including plasma inflammatory markers, serum and urinary advanced glycation (AGE) and lipoxidation (ALE) end-products (tertiary outcomes).

This trial will provide evidence for use of carnosine as a therapeutic intervention for PVD patients and, if positive, will have immediate clinical application.

DETAILED DESCRIPTION:
Peripheral vascular disease (PVD) has high prevalence of 10-15% in Australia and is caused by atherosclerotic occlusion of the arteries supplying the lower extremities which reduces blood flow and leads to intermittent claudication and critical limb ischaemia. No effective medication is currently available. Although surgical or endovascular revascularisation are available treatments, not all patients are suitable for the procedure, and grafts can fail, and dilated arteries can restenose. Structured exercise, both supervised and home-based, improves walking endurance in patients with PVD to a similar extent as revascularisation and effects are longer lasting but the pain associated with exercise is a major limitation. Therefore, there is a need to develop safe interventions synergistic with exercise that can prompt revascularisation and preserve limb viability.

Angiogenesis plays an essential role for recovery from critical limb ischaemia. Hypoxia inducible factor 1α (HIF1-α), a master regulator of angiogenic genes, has been implicated . Under normal conditions, HIF1-α is targeted for proteasomal degradation through the activity of prolyl hydroxylases (PHDs). PHDs require iron for their activity and their inactivation by metal chelators or pharmacological inhibitors stabilises HIF1-α and has been shown to improve blood flow in the ischaemic limb. However, metal chelators cannot be used as an intervention due to their toxicity.

Recent studies have shown that supplementation of carnosine (β-alanyl-L-histidine), a naturally occurring histidyl dipeptide in skeletal muscle with an excellent safety profile, improves exercise performance in athletes as well as in patients with chronic heart failure. The investigators and others have shown that carnosine supplementation also improves cardiometabolic risk factors. No clinical trial has yet to investigate whether carnosine improves walking endurance in patients with PVD. Carnosine has anti-inflammatory, antioxidative, anti-glycating and anti-atherosclerotic properties. It also has the ability to chelate metals, form conjugates with reactive aldehydes, and has lactate buffering capacity. In addition, carnosine has been found to be very effective in reducing ischaemia-reperfusion damage in several organs. Our preliminary results using a murine model of hind limb ischaemia (HLI) showed that administration of carnosine over 21 days increased HIF1-a and VEGF levels in the ischaemic muscle and improved tissue perfusion. Furthermore, mobilisation of pro-angiogenic endothelial progenitor cells (EPCs) and the ambulatory movement were increased in carnosine treated HLI mice compared to controls. The investigators propose a randomised clinical trial to investigate whether administration of carnosine for 6-month in addition to exercise could improve walking endurance and quality of life in patients with PVD compared to placebo and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age >=40or <80 years
* Clinical diagnosis Peripheral Vascular disease
* Rutherford Grade 1-3
* No significant kidney, cardiovascular, haematological, respiratory, gastrointestinal, or central nervous system disease, as well as no psychiatric disorders, no active cancer within the last five years; no presence of acute inflammation (by history, physical or laboratory examination)
* Intermittent claudication on treadmill between 30m and 200m
* Ankle Brachial index 0.6-1 at rest with minimum post exercise drop in ABI of 0.1

Exclusion Criteria:

* Age < 40 or > 80 years
* Pregnant or lactating
* Limb threatening ischaemia- Rutherford grades 4-6, manifested by ischaemic rest pain, ulceration, or gangrene; acute limb-threatening ischaemia
* lower limb surgical or endovascular interventions in the preceding 6 months
* planned lower limb endovascular or surgical intervention within the next 6 months on either limb
* taking medication for PVD (Cilostazol and Pentoxifylline)
* inability to complete the treadmill walking test for reasons other than claudication
* myocardial infarction within last 3 months
* deep vein thrombosis within 3 months
* estimated life expectancy < 1 year
* alcohol and illicit drug abuse.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
walking endurance | 6 months
  change in walking endurance (6-min walk test)

CONTACTS AND LOCATIONS:
Overall Officials: Barbora deCourten, MD,PHD,MPH, Principal Investigator — Monash University and Monash Health
Locations (1):
- Monash Centre for Health Research and Implementation, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No